CLINICAL TRIAL: NCT06672887
Title: Effectiveness, Cost-effectiveness, and Return on Investment of the Web-based MiLES Intervention Targeted at Employers, to Enhance Successful Return to Work of Employees With Cancer
Brief Title: Enhancing Successful Return to Work of Employees With Cancer, by Supporting Employers (MiLES Intervention)
Acronym: MiLES
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Cancer Society (Other); Re-turn (Unknown); Arbo Unie (Unknown)
Responsible Party: Principal Investigator, Michiel Greidanus, Postdoc researcher, Amsterdam UMC, location AMC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023.0524
Record Dates: First submitted 2024-10-25; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Neoplasm
Keywords: Cancer survivor; Employee with cancer; Employer; Return to work; Employment; Manager; Employee
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: A non-blinded RCT. The investigators will include employer-employee with cancer dyads, and will compare an intervention group, in which the employer will get access to the MiLES intervention, with a control group, in which both the employee and employer will receive care as usual.
Who Masked: Outcomes Assessor
Masking Description: Participants will not be blinded, as it was hard to devise a placebo intervention, and the standard care (no access to the MiLES intervention) was obviously different from the intervention (access to the MiLES intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Employers randomized to the intervention group will get a personal link to the MiLES intervention.
  Interventions: Other: MiLES
- Control group (No Intervention): The employees randomized to the control group will receive "care as usual" from their employer, as well as from their reintegration consultant or occupational physician. Their employer will not have access to the MiLES intervention during the study period. However, they will gain access for 6 months following a waiting-list period of 12 months.

INTERVENTIONS:
Other: MiLES — The MiLES intervention is an open access website, accessible via an URL, but not traceable through any online search engine during the study period. Tailored for specific preferences and needs of different employees with cancer, the MiLES intervention consists of interactive videos, conversation checklists, tips and information regarding RTW guidance of employees with cancer, and an overview of involved stakeholders and relevant legislation. The MiLES intervention intends to optimize the RTW support the employer provides to the employee with cancer by enhancing the willingness and ability to implement the employer actions. The MiLES intervention focuses for example on fostering effective communication between the employer and employee, while disregarding assumptions based on previous experiences.
  Arms: Intervention group

SUMMARY:
The objective of this randomized controlled trial (RCT) is to evaluate the effectiveness of the MiLES intervention targeted at employers, on successful return to work (RTW) of employees with cancer, compared to care as usual (CAU).

Secundary objectives are:

* To evaluate the cost-effectiveness and return-on-investment of the MiLES intervention on successful RTW and quality of life, compared to CAU.
* To evaluate the effectiveness of the MiLES intervention on several outcome measures on the level of the employee with cancer (time to RTW, quality of life, quality of working life, received work-related support, and satisfaction with work-related support), and the level of the employer (self-efficacy in providing RTW support, and satisfaction with the RTW process).

Participants will be 140 employer-employee with cancer dyads. All dyads will randomly be allocated to the intervention group, of which the employer will get unlimited access to the MiLES intervention, or to the control group in which CAU will be provided. The follow-up of this study will be 12 months.

Along with the RCT, a process evaluation using the UK Medical Research Council framework will also be conducted.

DETAILED DESCRIPTION:
The investigators will include 140 employer-employees with cancer dyads. The employees are diagnosed with cancer (<2 years earlier), aged 18-65 years, in paid employment with an employer, and currently fully or partly sick-listed (<2 years). The employer supports and guides the participating employee with cancer during the period of sick leave and RTW (e.g. as the direct supervisor or HR-manager).

Employers of dyads randomized to the intervention group will get unlimited access to the web-based MiLES intervention, aimed at enhancing the successful RTW of employees with cancer, by supporting employers. This intervention includes among others interactive video's, conversation checklists, and tips and information. Employers of dyads randomized to the control group will not get access to the MiLES intervention, thus dyads will get care as usual.

The primary outcome will be successful RTW, measured at the level of the employee. Secondary outcomes will include: current work situation (including time to RTW), quality of life and quality of working life, received work-related support, and satisfaction with work-related support. At the level of the employer, the secondary outcomes will include: self-efficacy in providing RTW support, and satisfaction with the RTW process. All outcomes will be assessed using questionnaires at baseline and at 3, 6 and 12 months of follow-up. Both the cost-effectiveness and the return on investment analysis will be conducted from the employers perspective. For the process evaluation, the UK MRC framework will be used.

ELIGIBILITY:
Inclusion criteria employees with cancer:

* Diagnosed with cancer <2 years earlier;
* Being of working age (between 18-65 years, considering the Dutch retirement age of 67 years, and the study's follow-up period of one year);
* In paid employment with an employer;
* Having either an occupational physician at the involved occupational health service or a reintegration consultant at the involved reintegration service (e.g. working for an organization that is affiliated with one of the settings of this study);
* Currently fully or partly sick-listed (<2 years);
* Able to understand and read Dutch for filling out questionnaires;
* Having already informed their employer about their diagnosis of cancer, or intending to do so;
* Not yet applied or planning to apply for an invalidity benefit under the WIA.

Inclusion criteria employers:

* Supports and guides the participating employee with cancer during the period of sick leave and RTW. For example, as the direct supervisor or HR-manager;
* Able to understand and read Dutch to be able to use the MiLES intervention and for filling out questionnaires;
* Not yet familiar with the MiLES intervention.

Exclusion Criteria:

- Employees with cancer and their employers must participate as a dyad. If one party in the dyad is unable or unwilling to participate, the other party cannot participate either.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Successful return to work (employee with cancer) | From enrollment to the end of the 12-month follow-up.
  The primary effect measure "successful RTW" is a combination of two components:
  1. Actual RTW: All employees will be asked about performed work activities in the past 4 weeks [yes/no]. This can be either their regular work activities or (temporarily) modified work activities.
  2. Successful RTW (14-items): Employees who have resumed work (actual RTW is answered by "yes") will also be asked about the extent to which they perceive their RTW as "successful", using the I-RTW_CS questionnaire.
  The I-RTW_CS is specifically developed as an RTW outcome measure that represents the perspectives of employees with cancer, with items that could be influenced by an employer.

SECONDARY OUTCOMES:
Current work situation (employee with cancer) | From enrollment to the end of the 12-month follow-up.
  Employees who have resumed work will be asked about their current work situation and since when they have returned to work (fully or partially). The questionnaire is self-developed and includes 9 items (e.g. time to RTW).
Quality of life (employee with cancer) | From enrollment to the end of the 12-month follow-up.
  The SF-12 questionnaire will be used to measure the perceived impact of health on a participant's everyday life (12 items).
Received work-related support from the employer (employee with cancer) | From enrollment to the end of the 12-month follow-up.
  Measured using self-developed questions, including the frequency of contact and its average duration (4-items).
Satisfaction with work-related support from their employer (employee with cancer) | From enrollment to the end of the 12-month follow-up.
  Measured on a self-developed 5-point Likert scale (1 item).
Quality of working life (employee with cancer) | From enrollment to the end of the 12-month follow-up.
  The Quality of Working Life Questionnaire for cancer survivors (QWLQ-CS) will be used to measure the experiences and perceptions at work over the past 4 weeks of employees who have resumed work.
Self-efficacy in providing return to work support (employer) | From enrollment to the end of the 12-month follow-up.
  Measured using an adapted version of the Competence scale of empowerment questionnaire (4 items).
Satisfaction with RTW process (employer) | From enrollment to the end of the 12-month follow-up.
  Measured on a self-developed 5-point Likert scale (1 item).

OTHER OUTCOMES:
Cost-effectiveness and return on investment | From enrollment to the end of the 12-month follow-up.
  The cost-effectiveness analysis and the return on investment analysis will be conducted from the employer's perspective, comparing the MiLES intervention with care as usual. They will be conducted for the primary outcome measure (i.e. successful RTW) and quality-adjusted life years (QALYs).

CONTACTS AND LOCATIONS:
Overall Officials: Sietske Tamminga, PhD, Principal Investigator — Amsterdam UMC, location AMC
Locations (5):
- Netherlands (5):
  - Arbo Unie, Arnhem
  - Arbo Unie, Dordrecht
  - Arbo Unie, Hengelo
  - Re-turn, Utrecht
  - Arbo Unie, Zeeland

IPD SHARING:
Plan to Share IPD: Undecided
Not yet determined

REFERENCES:
- [Derived] Mollet JM, Greidanus MA, Boot CRL, Vis C, van Dongen JM, de Boer AGEM, Tamminga SJ. Effectiveness, cost-effectiveness, and return on investment of the web-based MiLES intervention targeted at employers, to enhance successful return to work of employees with cancer: design of a randomized controlled trial. Trials. 2025 Oct 16;26(1):417. doi: 10.1186/s13063-025-09092-2. PMID 41102780